CLINICAL TRIAL: NCT05170113
Title: A Pilot, Randomized, Double-blind, Placebo-controlled, Parallel Design Study to Evaluate the Effectiveness and Safety of an Alpinia Galanga Formulation, Theacrine Formulation, and Caffeine Formulation on Fatigue, Mental Acuity, and Cognitive Health Among Overall Healthy Participants
Brief Title: Evaluate the Effectiveness and Safety of the Alpinia Galanga Formulation, Theacrine Formulation, and Caffeine Formulation on Fatigue, Mental Acuity, and Cognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: CL101
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Fatigue
Keywords: Energy; Fatigue; Tired; Sleep; Cognitive Health; Mental Acuity
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alpinia galanga formulation (Active Comparator): Alpinia galanga formulation capsule: Take one (1) capsule once daily at noon with 8 oz. (240 ml) of water for a 14-day dosing period
  Interventions: Dietary Supplement: Alpinia galanga formulation
- Theacrine formulation (Active Comparator): Theacrine formulation capsule: Take one (1) capsule once daily at noon with 8 oz. (240 ml) of water for a 14-day dosing period
  Interventions: Dietary Supplement: Theacrine formulation
- Caffeine formulation. (Active Comparator): Caffeine formulation capsule: Take one (1) capsules once daily at noon with 8 oz.(240 ml) of water for a 14-day dosing period
  Interventions: Dietary Supplement: Caffeine formulation
- Placebo (Placebo Comparator): Placebo capsule: Take one (1) capsule once daily at noon with 8 oz. (240 ml) of water for a 14-day dosing period
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpinia galanga formulation — Alpinia galanga formulation capsule- 1 capsule daily
  Arms: Alpinia galanga formulation
Dietary Supplement: Theacrine formulation — Theacrine formulation capsule- 1 capsule daily
  Arms: Theacrine formulation
Dietary Supplement: Caffeine formulation — Caffeine formulation capsule- I capsule daily
  Arms: Caffeine formulation.
Dietary Supplement: Placebo — Placebo capsule- 1 capsule daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of the Alpinia galanga formulation, Theacrine formulation, and Caffeine formulation on fatigue, mental acuity, and cognitive health among overall healthy participants

DETAILED DESCRIPTION:
This is a 4-arm pilot, double-blind, randomized, placebo-controlled, parallel design study. A total of 80 subjects (20 per treatment arm) will be enrolled in a randomly assigned sequence to receive either the Alpinia galanga formulation, Theacrine formulation, Caffeine formulation, or placebo in individuals and admit to experiencing occasional fatigue (tiredness) and would like more energy.

Participants will need to complete assessments and questionnaires.

The primary objective is the evaluation of the change in the response to the VAS-F (Visual Analogue Scale to Evaluate Fatigue Severity) relative to baseline. The secondary objective is the evaluation of the change in the responses to the BCAT-SF (Brief Cognitive Health Assessment Short Form), LSEQ (Leeds Sleep Evaluation Questionnaires), and SF-36 Health Survey (Short Form 36) compared to baseline.

Safety and tolerability will be evaluated through the receipt of documentation and responses from the telephone contacts/ emails per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 30-70 years of age
2. A body mass index (BMI) of 18.5 - 34.9
3. Admits to experiencing occasional fatigue (tiredness) and would like more energy
4. Has consumed no more than two cups of coffee or caffeinated beverage per day for seven or more days before Screening/baseline
5. Has personal access to and able to operate a smartphone, tablet, or computer with enough memory to accommodate additional application(s) and reliable internet service
6. Able to complete tests online with a computer
7. Able to print out and return documents by scan, email, or mail
8. Has regular daytime work hours or shifts, if employed (regular shift excludes night shift workers and those with rotating shifts)
9. Generally healthy and having no significant difficulty with digestion or absorption of food
10. Able to complete an Activity Log and Study Product Log daily
11. Has been generally weight stable for the past six months (give or take 6 lbs.)
12. Willing and able to give written informed consent
13. Clearly understands the procedures and study requirements
14. Willing and able to comply with all study procedures, as per protocol
15. Able to communicate, including reading, in English
16. Has not taken any nutritional supplements that may contain any of the components of the study products including Alpinia galanga, Theacrine or Caffeine for a minimum of 14 days before Screening/baseline

Exclusion Criteria:

1. Not having the basic skills needed to operate a smartphone, tablet, or computer
2. Unwilling to abstain from consuming more than two cups of coffee or caffeinated beverage/food per day and no caffeinated beverage/food after 10 am daily for the duration of the study
3. Having smoked any cigarette, electronic cigarette, cigar, or pipe, or used marijuana, any recreational drug or cannabidiol (CBD) in the past 30 days
4. Donated blood within the 30 days prior to Screening/baseline
5. Having participated in another study within 30 days before Screening/baseline
6. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
7. History of allergy or sensitivity to any component of the study products
8. Currently taking or having taken within the 30 days prior to Screening/baseline any medication(s) or supplement(s) which may have a stimulant effect in the judgment of the Study Investigator/Sub-investigator
9. Having been diagnosed, received medical treatment, or taking medication daily for any of the following medical condition(s):

   * Chronic fatigue syndrome
   * Fibromyalgia
   * Sleep disorder, including sleep apnea
10. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus or other endocrine disease
    * Eating disorder
    * Acute or chronic inflammatory disease or autoimmune disease
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke, or heart valve problem
    * Having a history of an abnormal electrocardiogram (ECG) unless permitted to proceed in the judgment of the Study Investigator/Sub-Investigator(s)
    * Gastrointestinal disease including gallbladder problems, gallstones, or biliary tract obstruction
    * Thyroid disease (unless on a stable dose of medication for 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Hypertension (unless on a stable dose of medication for 3 months before Screening/baseline and unlikely to change medication or dose during the study)
    * Neurologic condition/disease
    * Cancer (unless skin cancer other than melanoma which has been treated > 3 years before Screening/baseline)
    * Liver, pancreatic, and kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Other condition or medication use that would preclude participation in the study in the judgment of the Study Investigator/Sub-Investigator
11. Currently taking any medications or treatment for a psychiatric disorder (bipolar disorder, manic disorder, schizophrenia, apathetic [inherited] disorder), including antidepressant drugs, selective serotonin reuptake inhibitors (SSRIs), tricyclic and atypical antidepressants, benzodiazepines, CNS depressants, dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs), pentazocine, phenothiazines, and tramadol. These may preclude participation in the study depending on the judgment of the Study Investigator/Sub-Investigator
12. Currently taking or having taken within the 30 days before Screening/baseline any hormone replacement therapy (including DHEA, estrogen, progesterone, or testosterone; except those utilized as a method of birth control and which have been taken for > 3 months, with no anticipated change for the duration of the study). This may preclude participation in the study depending on the judgment of the Study Investigator/Sub-Investigator
13. Having had a surgical procedure or having an internal medical device which, in the judgment of the Study Investigator/Sub-Investigator, would preclude participation in the study
14. Currently consumes more than 7 standard alcoholic drinks per week for women and 14 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
15. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges, and tangelos for the study period
16. History of known or suspected substance abuse (e.g., alcohol, opiates, Benzodiazepines, or amphetamines)
17. Having any other circumstance that precludes study participation in the judgment of the Study Investigator/Sub-Investigator including use of other nutritional supplements, which will be evaluated on a case-by-case basis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
VAS-F (Visual Analogue Scale to Evaluate Fatigue Severity) | 14 Days
  Assessment of the mean change in the results of the VAS-F survey from baseline. This consists of 18 items relating to the subjective experience of fatigue with a Fatigue subscale and Energy subscale. The scores can range from 0-10 and the lower the score indicates a better outcome.

SECONDARY OUTCOMES:
BCAT-SF (Brief Cognitive Health Assessment Short Form) | 14 Days
  Assessment of the mean change in the results of the Brief Cognitive Assessment Tool (BCAT-SF) survey from baseline. It is a 6-item instrument with a score range of 0-21. The higher the score indicates a better outcome.

OTHER OUTCOMES:
LSEQ (Leeds Sleep Evaluation Questionnaires) | 14 Days
  Assessment of the mean change in the results of the Leeds Sleep Evaluation Questionnaire (LSEQ) survey from baseline. This questionnaire consists of ten self-rating questions related to four consecutive aspects of sleep (getting to sleep. quality of sleep, awakening from sleep and behavior following sleep). The total LSEQ socre can range from 0-100. The higher the total global LSEQ score indicates a better outcome.
SF-36 Health Survey (Short Form 36) | 14 Days
  Assessment of the mean change in the results of the Short Form-36 (SF-36) Health survey from baseline. This is a 36-item questionnaire that coversa eight domains including physiccal functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. The socres from each domain can range from 0-100, The higher the scores for each domain indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, PhD, Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alajmi MF, Mothana RA, Al-Rehaily AJ, Khaled JM. Antimycobacterial Activity and Safety Profile Assessment of Alpinia galanga and Tinospora cordifolia. Evid Based Complement Alternat Med. 2018 Jul 8;2018:2934583. doi: 10.1155/2018/2934583. eCollection 2018. PMID 30069222
- [Background] Alpinia. (2019, October 7). Natural medicines (database on the Internet). Somerville, MA: Therapeutic Research Center. Retrieved from https://naturalmedicines.therapeuticresearch.com/databases/food,-herbssupplements/professional.aspx?productid=276
- [Background] Bello ML, Walker AJ, McFadden BA, Sanders DJ, Arent SM. The effects of TeaCrine(R) and caffeine on endurance and cognitive performance during a simulated match in high-level soccer players. J Int Soc Sports Nutr. 2019 Apr 18;16(1):20. doi: 10.1186/s12970-019-0287-6. PMID 30999897
- [Background] Brice CF, Smith AP. Effects of caffeine on mood and performance: a study of realistic consumption. Psychopharmacology (Berl). 2002 Nov;164(2):188-92. doi: 10.1007/s00213-002-1175-2. Epub 2002 Sep 4. PMID 12404081
- [Background] Caffeine. (2020, January 6). Natural Medicines (database on the Internet). Somerville, MA: Therapeutic Research Center. Retrieved from https://naturalmedicines.therapeuticresearch.com/references.aspx?productid=979
- [Background] Carman AJ, Dacks PA, Lane RF, Shineman DW, Fillit HM. Current evidence for the use of coffee and caffeine to prevent age-related cognitive decline and Alzheimer's disease. J Nutr Health Aging. 2014 Apr;18(4):383-92. doi: 10.1007/s12603-014-0021-7. PMID 24676319
- [Background] Chudiwal, A., Jain, D., & Somani, R. (2010). Alpinia galanga Willd.-An overview on phytopharmacological properties. Indian Journal of Natural Products and Resources, 1(2), 143-149.
- [Background] Clewell A, Hirka G, Glavits R, Palmer PA, Endres JR, Murbach TS, Marx T, Pasics Szakonyine I. A 90-Day Oral Toxicological Evaluation of the Methylurate Purine Alkaloid Theacrine. J Toxicol. 2016;2016:6206859. doi: 10.1155/2016/6206859. Epub 2016 Aug 22. PMID 27635133
- [Background] Dallal, G. (2017, July 10). www.Randomization.com. Retrieved from Randomization.com: http://www.randomization.com
- [Background] Fredholm BB, Battig K, Holmen J, Nehlig A, Zvartau EE. Actions of caffeine in the brain with special reference to factors that contribute to its widespread use. Pharmacol Rev. 1999 Mar;51(1):83-133. No abstract available. PMID 10049999
- [Background] Ghosh S, Rangan L. Alpinia: the gold mine of future therapeutics. 3 Biotech. 2013 Jun;3(3):173-185. doi: 10.1007/s13205-012-0089-x. Epub 2012 Sep 18. PMID 28324376
- [Background] Haller CA, Jacob P 3rd, Benowitz NL. Pharmacology of ephedra alkaloids and caffeine after single-dose dietary supplement use. Clin Pharmacol Ther. 2002 Jun;71(6):421-32. doi: 10.1067/mcp.2002.124523. PMID 12087345
- [Background] Haskell CF, Kennedy DO, Wesnes KA, Scholey AB. Cognitive and mood improvements of caffeine in habitual consumers and habitual non-consumers of caffeine. Psychopharmacology (Berl). 2005 Jun;179(4):813-25. doi: 10.1007/s00213-004-2104-3. Epub 2005 Jan 28. PMID 15678363
- [Background] Taylor L, Mumford P, Roberts M, Hayward S, Mullins J, Urbina S, Wilborn C. Safety of TeaCrine(R), a non-habituating, naturally-occurring purine alkaloid over eight weeks of continuous use. J Int Soc Sports Nutr. 2016 Jan 13;13:2. doi: 10.1186/s12970-016-0113-3. eCollection 2016. PMID 26766930
- [Background] He H, Ma D, Crone LB, Butawan M, Meibohm B, Bloomer RJ, Yates CR. Assessment of the Drug-Drug Interaction Potential Between Theacrine and Caffeine in Humans. J Caffeine Res. 2017 Sep 1;7(3):95-102. doi: 10.1089/jcr.2017.0006. PMID 28875060
- [Background] Kamimori GH, McLellan TM, Tate CM, Voss DM, Niro P, Lieberman HR. Caffeine improves reaction time, vigilance and logical reasoning during extended periods with restricted opportunities for sleep. Psychopharmacology (Berl). 2015 Jun;232(12):2031-42. doi: 10.1007/s00213-014-3834-5. Epub 2014 Dec 21. PMID 25527035
- [Background] Kuhman DJ, Joyner KJ, Bloomer RJ. Cognitive Performance and Mood Following Ingestion of a Theacrine-Containing Dietary Supplement, Caffeine, or Placebo by Young Men and Women. Nutrients. 2015 Nov 19;7(11):9618-32. doi: 10.3390/nu7115484. PMID 26610558
- [Background] McLellan TM, Caldwell JA, Lieberman HR. A review of caffeine's effects on cognitive, physical and occupational performance. Neurosci Biobehav Rev. 2016 Dec;71:294-312. doi: 10.1016/j.neubiorev.2016.09.001. Epub 2016 Sep 6. PMID 27612937
- [Background] Institute of Medicine (US) Committee on Military Nutrition Research. Caffeine for the Sustainment of Mental Task Performance: Formulations for Military Operations. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK223802/ PMID 25057583
- [Background] Meredith SE, Juliano LM, Hughes JR, Griffiths RR. Caffeine Use Disorder: A Comprehensive Review and Research Agenda. J Caffeine Res. 2013 Sep;3(3):114-130. doi: 10.1089/jcr.2013.0016. PMID 24761279
- [Background] Nehlig A. Is caffeine a cognitive enhancer? J Alzheimers Dis. 2010;20 Suppl 1:S85-94. doi: 10.3233/JAD-2010-091315. PMID 20182035
- [Background] Office of New Drugs. (2005). Guidance for Industry Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. 1-37. Office of the Federal Register , National Archives and Record Administration.
- [Background] Qureshi S, Shah AH, Ageel AM. Toxicity studies on Alpinia galanga and Curcuma longa. Planta Med. 1992 Apr;58(2):124-7. doi: 10.1055/s-2006-961412. PMID 1529022
- [Background] Rosner, B. (n.d.). Hypothesis Testing: Two-Sample Inference-Estimation of Sample Size and Power for Comparing Two Means. In B. Rosner, Fundamentals of Biostatistics. Cengage Learning. Retrieved from www.stat.buc.ca: https://www.stat.ubc.ca/~rollin/stats/ssize/n2.html
- [Background] Saha S, Banerjee S. Central nervous system stimulant actions of Alpinia galanga (L.) rhizome: a preliminary study. Indian J Exp Biol. 2013 Oct;51(10):828-32. PMID 24266107
- [Background] Sebastiao AM, Ribeiro JA. Tuning and fine-tuning of synapses with adenosine. Curr Neuropharmacol. 2009 Sep;7(3):180-94. doi: 10.2174/157015909789152128. PMID 20190960
- [Background] Hanish Singh JC, Alagarsamy V, Diwan PV, Sathesh Kumar S, Nisha JC, Narsimha Reddy Y. Neuroprotective effect of Alpinia galanga (L.) fractions on Abeta(25-35) induced amnesia in mice. J Ethnopharmacol. 2011 Oct 31;138(1):85-91. doi: 10.1016/j.jep.2011.08.048. Epub 2011 Sep 1. PMID 21911048
- [Background] Sivanandan, S., & Pimple, S. (2018). Molecular Docking Studies of Alpinia galanga Phytoconstituents for Psychostimulant Activity. Advances in Biological Chemistry, 8(4),69-80
- [Background] Srivastava S, Mennemeier M, Pimple S. Effect of Alpinia galanga on Mental Alertness and Sustained Attention With or Without Caffeine: A Randomized Placebo-Controlled Study. J Am Coll Nutr. 2017 Nov-Dec;36(8):631-639. doi: 10.1080/07315724.2017.1342576. Epub 2017 Sep 14. PMID 28910196
- [Background] Srivastava, S., & Pimple, S. (2017). Effects of Cymbopogon Flexuosus, Alpinia Galanga, and Glycyrrhiza Glabra on attention: A randomized double-blind, placebo-controlled pilot study. BAOJ Nutrition, 3, 042.
- [Background] van Gelder BM, Buijsse B, Tijhuis M, Kalmijn S, Giampaoli S, Nissinen A, Kromhout D. Coffee consumption is inversely associated with cognitive decline in elderly European men: the FINE Study. Eur J Clin Nutr. 2007 Feb;61(2):226-32. doi: 10.1038/sj.ejcn.1602495. Epub 2006 Aug 16. PMID 16929246
- [Background] Wang Y, Yang X, Zheng X, Li J, Ye C, Song X. Theacrine, a purine alkaloid with anti-inflammatory and analgesic activities. Fitoterapia. 2010 Sep;81(6):627-31. doi: 10.1016/j.fitote.2010.03.008. Epub 2010 Mar 20. PMID 20227468
- [Background] Warburton DM. Effects of caffeine on cognition and mood without caffeine abstinence. Psychopharmacology (Berl). 1995 May;119(1):66-70. doi: 10.1007/BF02246055. PMID 7675951
- [Background] Wedick NM, Brennan AM, Sun Q, Hu FB, Mantzoros CS, van Dam RM. Effects of caffeinated and decaffeinated coffee on biological risk factors for type 2 diabetes: a randomized controlled trial. Nutr J. 2011 Sep 13;10:93. doi: 10.1186/1475-2891-10-93. PMID 21914162
- [Background] Zampelas A, Panagiotakos DB, Pitsavos C, Chrysohoou C, Stefanadis C. Associations between coffee consumption and inflammatory markers in healthy persons: the ATTICA study. Am J Clin Nutr. 2004 Oct;80(4):862-7. doi: 10.1093/ajcn/80.4.862. PMID 15447891
- [Background] Ziegenfuss TN, Habowski SM, Sandrock JE, Kedia AW, Kerksick CM, Lopez HL. A Two-Part Approach to Examine the Effects of Theacrine (TeaCrine(R)) Supplementation on Oxygen Consumption, Hemodynamic Responses, and Subjective Measures of Cognitive and Psychometric Parameters. J Diet Suppl. 2017 Jan 2;14(1):9-24. doi: 10.1080/19390211.2016.1178678. Epub 2016 May 10. PMID 27164220
- [Background] Zwyghuizen-Doorenbos A, Roehrs TA, Lipschutz L, Timms V, Roth T. Effects of caffeine on alertness. Psychopharmacology (Berl). 1990;100(1):36-9. doi: 10.1007/BF02245786. PMID 2296626